CLINICAL TRIAL: NCT06788444
Title: Efficacy of a Single Low Dose of Esketamine for Patients With Irritable Bowel Syndrome: Study Protocol for a Randomised Controlled Trial
Brief Title: Efficacy of Esketamine for Patients With Irritable Bowel Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, Director of Department of Day surgery and Pain Management, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY2024-414-02
Record Dates: First submitted 2025-01-22; First posted 2025-01-23 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable bowel syndrome; esketamine
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Esketamine

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Masking Description: Single (Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The esketamine group (Experimental): The propofol is administered until the patients loss of consciousness. Then 0.2 mg/kg esketamine is then administered by the anesthesiologist. After the administration of 0.2 mg/kg esketamine is completed, the endoscopist will begin the colonoscopic procedure.
  Interventions: Procedure: The colonoscopy; Drug: Esketamine
- The control group (Placebo Comparator): The propofol is administered until the patients loss of consciousness. Then normal saline is then administered by the anesthesiologist. After the administration of normal saline is completed, the endoscopist will begin the colonoscopic procedure.
  Interventions: Procedure: The colonoscopy

INTERVENTIONS:
Procedure: The colonoscopy — Both groups continued to receive the usual standard of gastroenterology care throughout the study period. The patients undergo preoperative preparation according to the requirements of colonoscopy. After entering the endoscopy room, the routine monitoring including electrocardiogram, heart rate, noninvasive blood pressure (BP), respiratory rate, and oxygen saturation (SpO2) are applied for patients. All monitoring data including HR, BP and SpO2 will be recorded at intervals of 3min. Safety assessments will be performed throughout the the research process. As a risk mitigation measure, esketamine should not be administered in patients with systolic blood pressure (SBP) > 140 mmHg or diastolic blood pressure (DBP) >90 mmHg prior to administration.
  After the right upper limb venous access is opened, the patients is placed in the left lateral position. The oxygen mask is placed near the patients' nose and oxygen is provided by the mask for 6L/min during the colonoscopy.
Drug: Esketamine — The propofol is administered until the patients loss of consciousness (loss of the eyelash refex). The 0.2 mg/kg esketamine is then administered by the anesthesiologist, but should be discontinued if the SBP ≥200 mmHg or the DBP ≥110 mmHg. After the administration of the 0.2 mg/kg esketamine is completed, the endoscopist will begin the colonoscopic procedure.
  Arms: The esketamine group

SUMMARY:
To explore the efficacy of a single low dose of esketamine for patients with irritable bowel syndrome (IBS).

DETAILED DESCRIPTION:
The investigators aim to investigate the efficacy of a single low dose of esketamine in patients with irritable bowel syndrome (IBS), and to explore the etiology of IBS and the effective and rapid treatment for this etiology.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 - 60 years;
2. American Society of Anesthesiologists (ASA) physical status of I - II;
3. Body Mass Index (BMI) of 15 - 30;
4. Scheduled for colonoscopy;
5. Positive screening results according to the Rome IV diagnostic criteria for IBS;
6. Patients who met Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for Anxiety disorder (ANXD) and/or major depressive disorder (MDD) .

Exclusion Criteria:

1. GastrointestinalTract (GI) bleeding;
2. Any organic lesions confirmed by clinical examination, laboratory examination or colonoscopy；
3. A previous diagnosis of colon cancer, infammatory bowel disease or coeliac disease;
4. A history of weight loss (at least 10%) within six months;
5. A history of abdominal surgery (other than hernia repair or appendectomy);
6. Participate in other clinical trials within 3 months;
7. Patients older than 55 years of age who have not undergone a colonoscopy in the past 5 years；
8. Mental disorder patients with severe personality disorder, active suicidal ideation and history of self-harm within 1 year;
9. Allergy or any contraindications to the drugs used in the study, such as severe cardiovascular disease, refractory hypertension, or hyperthyroidism;
10. Drinking more than 50 units (1 unit refers to 10ml of pure alcohol) per week;
11. Pregnancy or breastfeeding.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 552 (Estimated)
Dates: Start 2025-09-18 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The IBS Severity Scoring System (IBS-SSS) | At baseline and at 3 days, 1 week, 3 weeks, 6 weeks after colonoscopy
  The IBS Severity Scoring System (IBS-SSS) at baseline and at 6 weeks after colonoscopy, which incorporates five typical symptoms of IBS (intensity of abdominal pain, frequency of abdominal pain, intensity of bloating, dissatisfaction with bowel habits, associated interference with daily life) [54-56]. Each symptom score ranges from 0 to 100 and a higher score indicates a more severe symptoms of IBS. The parenteral symptoms incorporates nausea/vomiting, early satiety, heartburn, headache, backache, body aches, thigh pain, lethargy, excess wind, and urinary symptoms. Patients with IBS may be categorized according to IBS-SSS, which are asymptomatic (<75), mild (75-175), moderate (176-300), and severe (>300). A reduction of ≥50 points is considered clinical improvement.

SECONDARY OUTCOMES:
The IBS Quality of Life (IBS-QOL) questionnaire | At baseline and at 3 days, 1 week, 3 weeks, 6 weeks after colonoscopy
  The IBS Quality of Life (IBS-QOL) questionnaire at baseline and at 6 weeks after colonoscopy, which consists of 8 subscales (dysphoria, activity interference, personal image, health concerns, food avoidance, social reaction, sexuality, social relationship), with a total of 34 questions. Each subscale score ranges from 0 to 100 points. A higher score indicates a better quality of life.
The Bristol Stool Form (BSF) scale | At baseline and at 3 days, 1 week, 3 weeks, 6 weeks after colonoscopy
  The Bristol Stool Form (BSF) scale at baseline and at 6 weeks after colonoscopy, which is used to record the difference in proportions of the patient's daily bowel habits (hard stools, normal stools, and loose stools).
The Hospital Anxiety and Depression Scale (HADS) | At baseline and at 3 days, 1 week, 3 weeks, 6 weeks after colonoscopy,
  The Hospital Anxiety and Depression Scale (HADS) at baseline and at 6 weeks after colonoscopy, which consists of two sub-scales. Each sub-scale consists of 7 items and each item scored from 0 to 3. A higher score indicates more severe anxiety or depression. A score of 11 or above can indicate clinically significant anxiety or depression.
The Patient Health Questionnaire-12 Somatic Symptom (PHQ-12 SS) Score | At baseline and at 3 days, 1 week, 3 weeks, 6 weeks after colonoscopy
  The Patient Health Questionnaire-12 Somatic Symptom (PHQ-12 SS) Score at baseline and at 6 weeks after colonoscopy, which includes 12 extra-GI symptoms such as back pain, limb pain, and headache. A higher score indicates more severe somatization symptoms.
The respiratory and cardiovascular adverse events | At baseline and at 24 hours after colonoscopy
  The occurrence of the respiratory and cardiovascular adverse events such as tachycardia, elevated BP, hypotension, bradycardia and respiratory depression
The other adverse events | At baseline and at 24 hours after colonoscopy
  The occurrence of the other adverse events such as nausea, vomiting, dizziness, agitation, sedation and hallucinations.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Not yet decided

REFERENCES:
- [Derived] Sun Z, Jiang L, Xing Y, Luo F. Efficacy of a single low dose of esketamine for patients with irritable bowel syndrome: study protocol for a randomised controlled trial. BMJ Open. 2025 Jun 23;15(6):e099793. doi: 10.1136/bmjopen-2025-099793. PMID 40550724